CLINICAL TRIAL: NCT03219736
Title: A Randomized Controlled Trial of Non-Invasive Positive Airway Pressure in the Pediatric Emergency Department for the Treatment of Acute Asthma Exacerbations
Brief Title: NiPPV in the Treatment of Acute Asthma Exacerbations
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI could not get support for project. PI left UAMS
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NiPPV Asthma
Record Dates: First submitted 2014-07-02; First posted 2017-07-17 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-06

CONDITIONS: Bronchial Asthma; Status Asthmaticus
MeSH Terms: conditions — Asthma; Status Asthmaticus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Active Comparator): This group will receive all standard of care therapies as per the pediatric ED Asthma Severity Protocol. To summarize, all moderate and severe acute asthma exacerbations receive albuterol and atrovent continuous aerosols, oral or intravenous steroids and intravenous magnesium sulfate. At the discretion of the treating physician, the patient may also receive subcutaneous terbutaline or epinephrine
  Interventions: Procedure: Standard of Care therapies; Procedure: Routine Respiratory Care
- NiPPV (Active Comparator): This group will receive all standard of care therapies as per the pediatric ED Asthma Severity Protocol. All nebulized treatments will be given via the NIPPV/BiPAP machine (EnVe Ventilator). Optimal settings for each participant should be achieved within 20 minutes of initiation of NiPPV. Pediatric asthma scores will continue to be recorded at least every hour or with every physician suggested NIPPV ventilator setting change for an 8 hour period. Furthermore, the NIPPV machine in conjunction with NM3 volumetric end tidal CO2 monitoring will record ventilatory data in this NIPPV/BiPAP group and will be compared to other study groups. The subjects will remain in the study for minimum of 4 hrs NIPPV therapy and total of 8 hours.
  Interventions: Device: NiPPV Therapy; Procedure: Routine Respiratory Care

INTERVENTIONS:
Procedure: Standard of Care therapies — If at any point during the treatment it is deemed medically necessary by the treating PED attending that a subject from the control arm (Group 1) requires an escalation of therapy, they may be moved from the group to the NIPPV/BiPAP group (Group 2) or be removed from the study (i.e. if intubated).
  Arms: Control
Device: NiPPV Therapy — If at any point during the treatment it is deemed medically necessary by the treating PED attending that a subject from a NIPPV/BiPAP group (Group 2) is not tolerating NIPPV they may be removed from the study. Patients may not tolerate NIPPV due to agitation, vomiting or need for escalation of care.
  Other Names: Bipap Therapy, Servo i ventilator by Maquet
  Arms: NiPPV
Procedure: Routine Respiratory Care — It may be up to the treating physicians discretion to treat patient with other medications that are currently used to treat severe asthma exacerbations, such as Epinephrine and Terbutaline

SUMMARY:
Study Summary:

Title: A Randomized Controlled Trial of Noninvasive Positive Airway Pressure in the Pediatric Emergency Department for the Treatment of Acute Asthma Exacerbations

Principal Investigator: Thomas J. Abramo, MD

Hypothesis: For acute moderate to severe pediatric asthma exacerbations the use of NIPPV/BiPAP, in conjunction with current standard of care therapies, will lead to a more rapid improvement in patient ventilation, faster resolution of respiratory distress and result in improved ventilatory parameters, secondary outcomes and pediatric asthma scores.

Study Design: Prospective, randomized controlled trial

Study Duration: This study will be conducted over a 36 month period.

Sample Size: 240 subjects

Population: Children ages 2-17 years of age presenting to the ED with Acute asthma exacerbation and a Pediatric Asthma Score (PAS) ≥ 8.

Synopsis: Eligible subjects will be randomized to either a control group or study groups. The study groups will be either a NIPPV/BiPAP group. The subjects in the study groups will continue to receive all standard of care therapies per the asthma severity protocols. All nebulized therapies will be given through the NIPPV circuit. Patients will be assessed by the pediatric asthma score (PAS), measured respiratory parameters, volumetric end tidal carbon dioxide monitoring and measured cardiac parameters.

Objectives: A. Evaluate if the use of NIPPV/BiPAP in conjunction with traditional inhaled beta-agonists improves the outcome in pediatric patients with acute moderate to severe asthma in the acute setting.

B. Describe the physiology of NIPPV/BiPAP by measuring cardiac parameters in children randomized to a NIPPV group.

C. Monitor safety of NIPPV/BiPAP use for acute asthma exacerbations in children.

Safety A.: The study must be IRB approved.

B.: Appropriate consent and assent documents will be obtained prior to enrolling the subject in the study.

C.: A clear safety plan including DSMB will be established to monitor for adverse events.

D.: Confidentiality will be ensured for all subjects enrolled in the study.

DETAILED DESCRIPTION:
This study is a prospective and randomized clinical trial to investigate the utility of BiPAP therapy for the pediatric patient in an acute moderate to severe asthma exacerbation. The study will be conducted in the pediatric emergency department at Arkansas Children's Hospital. Patients between 2-17 years old will be identified to participate based on the past medical history, history of present illness and PAS and the consent process will begin immediately. All patients will be started on standard of care therapies including continuous albuterol and atrovent aerosols, intravenous corticosteroids, intravenous magnesium sulfate and a normal saline fluid bolus. Additional therapies with subcutaneous epinephrine or terbutaline will be given at the discretion of the treating physician in the first 20 minutes. Further escalation of asthma therapy, for example administration of IV bronchodilators, ketamine, terbutaline and/or epinephrine will be at the discretion of the treating physician. The history of present illness, past medical history, triage information and initial physical exam information will be collected by the study investigator in the first hour and marked on the data sheet.

Once consented, participants will be randomized to one of two groups by selection of an opaque folder by the study investigator. A PAS will be assigned at 1 hour after only having received traditional standard of care therapies and before placing the subject on the therapy determined by the randomization. If the child receives a score of 7 or less, he/she will not be placed on NIPPV; however, they will be analyzed in this group based on intention to treat.

i. Group #1: This group will receive all standard of care therapies as per the pediatric ED Asthma Severity Protocol. Will be referred to as the control group.

ii. Group #2: This group will receive all standard of care therapies as per the pediatric ED Asthma Severity Protocol. All nebulized treatments will be given via the NIPPV/BiPAP machine via the Servo i Ventilator. The treating PED Attending and treating PED respiratory therapist will be blinded to the BiPAP/NIPPV settings during the study period. The PED clinical trial research assistant and in conjunction with one of the study investigators will adjust the BiPAP settings in concert with the treating physician. The discussion will be about either increasing or decreasing the IPAP or EPAP not the true number changes to keep it blinded, will be as follows: The inspiratory positive airway pressure (IPAP) will be started at 10 cm H2O for all patients. The patient will be observed clinically by a PED respiratory therapist in conjunction with the treating pediatric ED attending and/or fellow. The IPAP will be increased as needed by 2 cm H2O up to a maximum IPAP of 16 cm H2O for patients 2-6 years of age, 20 cm H2O for patients 7-12 years of age, and 24 cm H2O for patients older than 12 years. The expiratory positive airway pressure (EPAP) will be set at 5 cm H2O. If the IPAP settings are maximized based on age and the respiratory distress score continues to be 5 or greater, the EPAP can be increased by 1 cm H2O to a maximum of 8 cm H2O for all patients less than 12 years and 10 cm H2O for all patients older than 12 years. The I:E setting will be 1.75 seconds. Optimal settings for each participant should be achieved within 20 minutes of initiation of BiPAP and respiratory distress scores should recorded at least every 5 minutes or with every BiPAP settings change during this period. Pediatric asthma scores will continue to be recorded at least every 30 minutes or with every physician suggested NIPPV ventilator setting change for an 8 hour period. Furthermore, the NIPPV ventilator, Servo i ventilator, has volumetric end tidal CO2 monitoring capabilities and will record ventilatory data in this NIPPV/BiPAP group and will be compared to other study groups.

The subjects will remain in the study for minimum of 4 hrs NIPPV therapy and total of 8 hours unless clinically still needing the NIPPV therapy. The first hour they will all receive the same standard therapies, followed by 7 hours of the therapies from the group in which they were randomized. Each 30 minutes in the study, the subject will be assessed by treating PED/PICU attending as to whether to continue the patient on the study arm, switch to a rescue arm or discontinue the patient from the study. This reassessment will be facilitated by the study investigator via a direct discussion with the treating attending physician. Furthermore, every 30 minutes the treating RT, treating PED attending or fellow, or study investigator will perform a PAS. Based on the PAS, the treating PED attending will be asked if patient needs further adjustment of the EnVe or continue present therapy. Once a subject in the NIPPV arm reaches a PAS of less than or equal to 7, the NIPPV settings may be weaned per the ACH PED NIPPV/BiPAP weaning protocol.

i. Rescue Arm A: If at any point during the treatment it is deemed medically necessary by the treating PED attending that a subject from the control arm, Group 1, requires an escalation of therapy, they may be moved from the group to the NIPPV/BiPAP group, Group 2, or be removed from the study i.e. if intubated.

ii. Rescue Arm B: If at any point during the treatment it is deemed medically necessary by the treating PED attending that a subject from a NIPPV/BiPAP group,Group 2, is not tolerating NIPPV they may be removed from the study. Patients may not tolerate NIPPV due to agitation, vomiting or need for escalation of care.

Additionally, in an attempt to better understand the physiology of NIPPV/BiPAP parameters of cardiac output, aortic flow and pulmonary flow, will be measured using the USCOM. This will assist us in understanding the physiological effects of the setting choices.

Subjects in Group 2 will be kept on the NIPPV machine for 4 hours minimum, unless the PED or PICU treating attending deems the patient has dramatically improved to take off the machine. The study investigator will collect information regarding medications given and any complications. At the end of the 8 hour study period, a PAS score will be calculated, and the study investigator will ask the PED or PICU treating attending whether to continue present therapy or switch to another therapy.

After the study time has completed, the study investigator will collect information such as PED/PICU diagnosis, disposition from PED/PICU and related information based on disposition, length of hospital stay and 72 hour returns from PED and mark it on the data sheet.

VII. Selection and enrollment of subjects

Inclusion criteria

2-17 years old For subjects 3 years and older, a known history of asthma as diagnosed by the PCP or per the ACH problem list For children ages 2-3 years, four or more episodes of wheezing in the past year that lasted more than 1 day and affected sleep AND one of the following: parental history of asthma, a physician diagnosis of atopic dermatitis, or evidence of sensitization to aeroallergens Acute asthma exacerbation Pediatric Asthma Score (PAS) ≥ 8 Parents willing and able to sign consent Children over the age of 6 willing to provide assent

Exclusion criteria

History of congenital heart disease, chronic respiratory disease including bronchopulmonary dysplasia, cystic fibrosis, pulmonary hypertension or any chronic lung disease other than asthma History of sickle cell disease Recently diagnosed pneumonia Current tracheostomy, on home ventilator or home oxygen requirement Recent diabetic ketoacidosis Requiring immediate intubation Weight less than 5 kilograms Any contraindication to BiPAP use including altered mental status, recent bowel surgery, intractable vomiting, inability to protect airway A history of prematurity of ≤ 30 weeks gestation

N/A

ELIGIBILITY:
Inclusion Criteria:

* 2-17 years old
* For subjects 3 years and older, a known history of asthma as diagnosed by the PCP or per the ACH problem list
* For children ages 2-3 years, four or more episodes of wheezing in the past year that lasted more than 1 day and affected sleep AND one of the following:

  * parental history of asthma, a physician diagnosis of atopic dermatitis, or evidence of sensitization to aeroallergens
* Acute asthma exacerbation
* Pediatric Asthma Score (PAS) ≥ 8
* Parents willing and able to sign consent
* Children over the age of 6 willing to provide assent

Exclusion Criteria:

* History of congenital heart disease, chronic respiratory disease including bronchopulmonary dysplasia, cystic fibrosis, pulmonary hypertension or any chronic lung disease other than asthma
* History of sickle cell disease
* Recently diagnosed pneumonia
* Current tracheostomy, on home ventilator or home oxygen requirement Recent diabetic ketoacidosis
* Requiring immediate intubation

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Decrease in the Pediatric Asthma Score within the designated time frame. | Every hour for a total of 8 hours
  The Research coordinator or Respiratory Therapist will measure a PAS every hour for a total of 8 hours with the goal of lowering the PAS

SECONDARY OUTCOMES:
Time to decrease PAS to less than 4 within 8 hours of initiation of NiPPV/Bipap | 8 hours
  The goal of the treatment strategy is to lower the PAS to less than 4 so that the patient may be transitioned from the NiPPV/Bipap to standard oxygen therapy for the treatment of an exacerbation of their asthma
Measurement of volumetric end tidal CO2 trend with the NICO2® Respiratory volumetric capnography CO2 monitors. | 8 hours
  The goal of the therapy is to be able to reduce the amount of inspiratory pressure the patient receives as their disease process improves. We hope to measure this with the end-tidal CO2 device. When the exhaled CO2 trends down we hope to reduce the inspiratory pressure the patient is receiving via NiPPV/BiPAP
Analysis of flow loops captured by the NIPPV device. | 8 hours
  By the Respiratory therapist and physician examining the flow volume loops from the patient data, we hope to capture the time that the patients lungs have seen a reduction in bronchospasms
Changes in individual pulmonary parameters: respiratory rate | 8 hours
  By adding NiPPV/Bipap to the patient to increase their inspiratory pressure while receiving their respiratory medications, we hope to be able to get the medications to the lower airways faster to help patient recover faster from asthma exacerbation which will hopefully reduce patient's length of stay in the hospital
Changes in individual pulmonary parameters: Oxygen requirement | 8 hours
  By adding NiPPV/Bipap to the patient to increase their inspiratory pressure while receiving their respiratory medications, we hope to be able to get the medications to the lower airways faster to help patient recover faster from asthma exacerbation which will hopefully reduce patient's length of stay in the hospital
Changes in individual pulmonary parameters: Oxygen saturations | 8 hours
  By adding NiPPV/Bipap to the patient to increase their inspiratory pressure while receiving their respiratory medications, we hope to be able to get the medications to the lower airways faster to help patient recover faster from asthma exacerbation which will hopefully reduce patient's length of stay in the hospital
Changes in cardiac parameters as measured by the USCOM, to include intubation rates, decrease length of hospital stay, limited need for additional treatments, ICU admission, barotrauma effects, and death. | 8 hours
  We hope to show improvements in Cardiac output measurements from the start of therapy until after treatment has been discontinued. We hope to show in increase in cardiac output due to the decrease in air trapping that is caused when a patient is undergoing an asthma exacerbation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Abramo, MD, Principal Investigator — UAMS/ACH
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States